CLINICAL TRIAL: NCT02585024
Title: Cytisine as a Smoking Cessation Agent: Improving Adherence Through a Better Understanding of Pharmacokinetics and Dose Response
Brief Title: Cytisine Pharmacokinetics and Dose Response (C-DRAKS 3 and C-DRAKS 4)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor, University of Auckland, New Zealand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AMRF reference 1 1 15 011
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
Keywords: smoking; cytisine; Pharmacokinetics
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1.5 mg cytisine (Experimental): 1.5 mg cytisine given as a single dose
  Interventions: Drug: Cytisine
- 3 mg cytisine (Experimental): 3 mg cytisine given as a single dose
  Interventions: Drug: Cytisine
- 4.5 mg cytisine (Experimental): 4.5 mg cytisine given as a single dose
  Interventions: Drug: Cytisine
- 1.5 mg cytisine six times a day (Experimental): 1.5 mg (1 capsule) is given six times a day (0, 2, 4, 6, 8 and 10 hours) for 5 days
  Interventions: Drug: Cytisine
- 3 mg cytisine three times a day (Experimental): 3 mg (2 capsules) are given three times a day (0, 4 and 8 hours) for 5 days
  Interventions: Drug: Cytisine
- 4.5 mg cytisine two times a day (Experimental): 4.5 mg (3 capsules) are given two times a day (0 and 6 hours) for 5 days
  Interventions: Drug: Cytisine

INTERVENTIONS:
Drug: Cytisine
  Other Names: Cytisine, Desmoxan

SUMMARY:
A number of pharmacotherapies are available for smoking cessation in New Zealand including nicotine replacement therapy, bupropion, an antidepressant medication and varenicline. Of these, varenicline is the most effective, but also the most expensive. Varenicline acts like nicotine and stimulates nicotine receptors in the brain, but to a lesser extent, and simultaneously block nicotine binding to its receptors and thus reduces the rewarding effects of cigarette smoking. Cytisine (Tabex® and Desmoxan®) is a plant alkaloid and also acts in a similar way to varenicline but is significantly cheaper. It has been used for more than 50 years in some parts of eastern and central Europe as an aid to quit smoking, but is not approved for use in many countries such as New Zealand, Australia, the UK or the US. Randomised, placebo-controlled trials have shown that cytisine is more effective than placebo and nicotine replacement therapy (NRT)for smoking cessation. However there is a paucity of pre-clinical data on cytisine. In particular, there are limited data on the pharmacokinetic and the dose response characteristics of cytisine. Furthermore, the current dosing regimen recommended by the manufacturer is complex and has no clear basis in empirical research.

Complexity of dosing has been shown to be a key factor in determining adherence. Therefore, a simpler regimen would likely maximise the effectiveness of treatment through improved adherence to the treatment regimen. The investigators therefore propose to undertake two studies to investigate the influence of dose, dosing frequency and dosing duration on the pharmacokinetics and tolerability of cytisine and cigarette craving in smokers.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age,
* be able to provide written consent,
* have no significant medical or psychiatric disorder (see below under exclusion criteria)
* smoke at least 10 cigarettes a day

Exclusion Criteria:

* they are pregnant or breastfeeding,
* they are current users of NRT products,
* they are current users of non-NRT smoking cessation therapies (e.g. bupropion [Zyban®], clonidine, nortriptyline, or varenicline [Champix®]),
* they are enrolled in another smoking cessation programme (concurrent referral to a face-to-face provider from Quitline is acceptable) or other cessation study
* they have had a heart attack, stroke, or severe angina within the past three months,
* they have uncontrolled high blood pressure (> 150 mmHg systolic, > 100 mmHg diastolic),
* they have phaeochromocytoma,
* they have been diagnosed with epilepsy
* they suffer from significant mental health problems
* they have severe renal impairment
* they are taking medications which are significantly affected by cessation of smoking (e.g. warfarin, olanzapine, clozapine, therophylline, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Exposure (AUC) | Arms 1-3: 24 hours; Arms 4-6: 24 hours, and up to Day 5
  Plasma cytisine concentrations will be measured in all groups for 24 hours. For Arms 4-6, we will continue to take blood samples to measure cytisine concentrations throughout the dosing period (Days 1-5). Days 3-5: one blood sample will be taken before the first dose for the day. On Day 5 an extra blood sample will be taken at 7.5 hours post the first dose for that day.

SECONDARY OUTCOMES:
Nicotine and cotinine concentrations | Arms 1-3: 24 hours; Arms 4-6: 24 hours, and up to Day 5
  Plasma nicotine and cotinine concentrations will be measured along with cytisine concentrations (from the same plasma samples)
Craving for cigarettes | Arms 1-3: 0, 1, 2, 4, 6, 8, 10 and 24 hours. Arms 4-6: 0, 2, 4 ,6, 8, 10, 24 hours; once on Days 3- 5
  The brief Questionnaire on Smoking Urges will be administered
Blood pressure | Arms: 1-3: 0, 1, 2, 4, 6, 8, 10, 24 hours. Arms 4-6: 0, 2, 4, 6, 8, 10, 24 hours; once on Days 3- 5
  Systolic and diastolic blood pressure (mm Hg) will be measured with a blood pressure monitor
Heart rate | Arms: 1-3: 0, 1, 2, 4, 6, 8, 10, 24 hours. Arms 4-6: 0, 2, 4, 6, 8, 10, 24 hours; once on Days 3- 5
  Heart rate (beats per minute) will be simultaneously measured with blood pressure using a blood pressure monitor
Respiratory rate | Arms: 1-3: 0, 1, 2, 4, 6, 8, 10, 24 hours. Arms 4-6: 0, 2, 4, 6, 8, 10, 24 hours; once on Days 3- 5
  Respiratory rate (breaths per minute) will be measured along with blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Soo Hee Jeong, Phd, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Soo Hee Jeong, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong SH, Sheridan J, Bullen C, Newcombe D, Walker N, Tingle M. Ascending single dose pharmacokinetics of cytisine in healthy adult smokers. Xenobiotica. 2019 Nov;49(11):1332-1337. doi: 10.1080/00498254.2018.1557760. Epub 2019 Jun 19. PMID 30526213